CLINICAL TRIAL: NCT06952751
Title: Optimization of the Isolation Protocol for Extracellular Vesicles (EVs) From Human Follicular Fluid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2024-0419; G096624N (Other Grant/Funding Number: FWO)
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Extracellular Vesicles
Keywords: Extracellular vesicles; Isolation
MeSH Terms: interventions — Chromatography, Gel

STUDY DESIGN:
Intervention Model Description: All collections of follicular fluid will be divided to test all three isolation methods under investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Intervention group
  Interventions: Other: Differential ultracentrifugation; Other: OptiPrep™ density gradient ultracentrifugation; Other: Size-exclusion chromatography; Other: Combined techniques

INTERVENTIONS:
Other: Differential ultracentrifugation — Differential ultracentrifugation
Other: OptiPrep™ density gradient ultracentrifugation — OptiPrep™ density gradient ultracentrifugation
Other: Size-exclusion chromatography — Size-exclusion chromatography
Other: Combined techniques — Combined techniques

SUMMARY:
Background: Extracellular vesicles (EVs) are membrane-bound vesicles found in all biological fluids, containing various regulatory molecules, including microRNAs (miRNAs). It has been suggested that the EVs in human follicular fluid (the fluid surrounding the oocyte within the ovary) play a crucial role in oocyte development through these miRNAs. However, several methods exist for isolating these EVs from follicular fluid. Before further research can be conducted on the pathophysiology and potential diagnostic and therapeutic applications of these EVs and their content, the optimal isolation technique must be determined for future studies.

Each method has its advantages and disadvantages, and the purity and efficiency may vary between species and different biological fluids. There are only a limited number of studies comparing the various techniques for application in human follicular fluid.

Objective: This study will compare the three most commonly used techniques for isolating EVs: size-based, sedimentation-based (differential ultracentrifugation), and buoyancy-based isolation techniques.

Methodology:

In this prospective study, follicular fluid will be collected from four patients undergoing transvaginal oocyte retrieval following ovarian stimulation at Ghent University Hospital. Patients over 40 years of age or with endometriosis, adenomyosis, or PCOS (polycystic ovarian syndrome) will not be included in this study. During the oocyte retrieval procedure, follicular fluid will be collected from 2-4 oocytes per patient. Since follicular fluid is not used in the patient's treatment (residual material), it does not affect the treatment.

After collection, the three isolation techniques will be applied to each sample. The techniques will be compared in terms of purity (absence of contamination) and efficiency (EV concentration) using transmission electron microscopy, nanoparticle tracking analysis, and western blotting.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for an oocyte retrieval at Ghent University Hospital.

Exclusion Criteria:

* Diagnosis of endometriosis/adenomyosis
* Diagnosis of PCOS (Polycystic Ovary Syndrome)
* Macroscopic blood contamination at oocyte retrieval

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Purety | 3 months
  Purety of EV isolation

SECONDARY OUTCOMES:
Efficiency | 3 months
  Efficiency in terms of number of particles
RNA efficiency | 6 months
  Efficiency in terms of RIN scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No